CLINICAL TRIAL: NCT02944162
Title: Clinical Investigation of Chimeric CD(Cluster of Differentiation)33 Antigen Receptor-modified NK92 Cells in Relapsed and/or Refractory Acute Myeloid Leukemias
Brief Title: CAR-pNK Cell Immunotherapy for Relapsed/Refractory CD33+ AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Hefei (Other); Hefei Binhu Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-0332
Record Dates: First submitted 2016-10-23; First posted 2016-10-25 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myelogenous Leukemia; Acute Myeloid Leukemia; Acute Myeloid Leukemia With Maturation; Acute Myeloid Leukemia Without Maturation; ANLL
Keywords: AML; CD33; CAR-NK
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sensitivity and Specificity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-NK Cell immunotherapy (Experimental): Enrolled patients will receive CAR-NK cells immunotherapy with a novel specific chimeric antigen receptor targeting CD33 antigen by infusion.
  Interventions: Biological: anti-CD33 CAR-NK cells

INTERVENTIONS:
Biological: anti-CD33 CAR-NK cells — The allogeneic NK cells (NK-92 cell line for clinical use) are engineered to contain anti-CD33 attached to TCRzeta, CD28 and 4-1BB signaling domains. These modified cells are called chimeric antigen receptor NK cells with specificity for CD33.
  Other Names: Chimeric antigen receptor NK92 cells with specificity for CD33

SUMMARY:
The purpose of this clinical trial is to study genetically engineered NK92 cell therapy in treating patients with CD33 positive acute myeloid leukemias that is relapsed (after stem cell transplantation or intensive chemotherapy) or refractory to further chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Determine the safety and feasibility of the chimeric antigen receptor NK92 cells transduced with the anti-CD33 vector (referred to as anti-CD33 CAR-NK cells).

SECONDARY OBJECTIVES:

I. For patients with detectable disease, measure anti-leukemia response due to anti-CD33 CAR-NK cell infusions.

II. For patients with stored or accessible leukemia blasts, determine leukemia cell killing by anti-CD33 CAR-NK in vitro.

III. Determine if cellular or humoral host immunity develops against the murine anti-CD33.

OUTLINE: Patients are assigned to 1 group according to order of enrollment.

Patients receive anti-CD33 CAR-NK (coupled with CD28, CD137 and CD3 zeta signalling domains) vector-transduced NK92 cell line on days 0,3, and 5 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with CD33+ acute myeloid leukemia in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (>12 weeks to < 2 year survival) with currently available therapies will be enrolled.
2. CD33+ acute myeloid leukemia CR (complete remission) can not be achieved after at least 2 prior combination chemotherapy regimens.
3. AML in CR2 or CR3 and not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor.
4. Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year).
5. Relapsed after prior autologous or allogenic SCT. AML patients with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT.
6. Residual disease after primary therapy and not eligible for autologous SCT.
7. All of those patients must also meet the following criteria:

Expected survival > 12 weeks. Creatinine < 2.5 mg/dl ALT(alanine aminotransferase)/AST (aspartate aminotransferase)< 3x normal Bilirubin < 2.0 mg/dl Any relapse after prior SCT will make patient eligible regardless of other prior therapy.

Adequate venous access for apheresis, and no other contraindications for leukapheresis.

Ability to give informed consent.

Exclusion Criteria:

1. Pregnant or nursing women may not participate.
2. Active HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at the time of screening.
3. Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
4. History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.
5. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
6. The existence of unstable or active ulcers or gastrointestinal bleeding.
7. Patients need anticoagulant therapy (such as warfarin or heparin).
8. Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the anti-CD33 CAR-NK cells | One year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Objective Response Rate | Up to one year
  Anti-leukemia responses to anti-CD33 CAR-NK cell infusions

CONTACTS AND LOCATIONS:
Locations (1):
- PersonGen BioTherapeutics (Suzhou) Co., Ltd., Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
(1) The use of a controlled access approach, using a transparent and robust system to review requests and provide secure data access; (2) Seeking consent for sharing IPD from trial participants in all future clinical trials with adequate assurance that patient privacy and confidentiality can be maintained; and (3) Establishing an approach to resource the sharing of IPD which would include support from trial funders, sponsor organisations and users of IPD.

REFERENCES:
- [Derived] Del Zotto G, Marcenaro E, Vacca P, Sivori S, Pende D, Della Chiesa M, Moretta F, Ingegnere T, Mingari MC, Moretta A, Moretta L. Markers and function of human NK cells in normal and pathological conditions. Cytometry B Clin Cytom. 2017 Mar;92(2):100-114. doi: 10.1002/cyto.b.21508. Epub 2017 Feb 12. PMID 28054442